CLINICAL TRIAL: NCT00567125
Title: A Comparative Study of Angiogenic and Cytokine Responses After Laparoscopic Cholecystectomy Performed With Standard-Pressure and Low-Pressure Pneumoperitoneum
Brief Title: Comparison of Systemic Response After Laparoscopies Performed With Standard and Low-Pressure Pneumoperitoneum
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Maciejewski Ryszard, MD, PhD, Medical University of Lublin
Other Study IDs: PW 205; PW 205/07
Record Dates: First submitted 2007-12-01; First posted 2007-12-04 (Estimated); Last update posted 2007-12-04 (Estimated); Status verified 2007-12

CONDITIONS: Laparoscopy.
Keywords: low-pressure pneumoperitoneum; laparoscopy; cytokines; VEGF-A; endostatin

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- I: Patients with cholelithiasis operated on using standard laparoscopy method
- II: Patients with cholelithiasis operated on using low-pressure CO2 pneumoperitoneum laparoscopy

SUMMARY:
The purpose of the study was the comparative assessment of the influence of low and standard pressure CO2 pneumoperitoneum on the systemic inflammatory and angiogenic responses during the postoperative period after laparoscopic management of cholelithiasis.

DETAILED DESCRIPTION:
Objective: The purpose of the study was to access the influence of low pressure CO2 pneumoperitoneum on the inflammatory and angiogenic responses during the postoperative period after laparoscopy. Summary background data: Surgical procedures enhance production of pro- and anti-inflammatory cytokines and angiogenic factors that play a pivotal role in the immunological response to surgical trauma and take part in the pathogenesis of tumor growth and adhesions formation. Methods: Study group consisted of 40 patients, operated on due to cholelithiasis using standard- (n=20) and low-pressure (n=20) CO2 pneumoperitoneum. Serum concentration of IL-6, IL-8, IL-10, VEGF-A and endostatin were measured before the surgeries and thereafter at 6, 24 and 48h with commercially available ELISA assays. Results: Concentrations of IL-6 increased significantly after the operations in both groups. No differences were observed between the groups in regards to IL-6, IL-8 and IL-10 levels. Concentrations of VEGF-A measured at 6 and 48h were significantly lower in patients who underwent laparoscopies performed with low pressure pneumoperitoneum. No significant variations were observed in endostatin serum concentration. Concentrations of the studied parameters were not influenced by the duration of surgeries, age, gender, or BMI of the patients. Conclusions: The results obtained in our study do not show any significant differences between studied operative procedures with regards to systemic inflammatory response. Changes in the concentrations of VEGF-A and endostatin observed in the studied population may suggest this technique to be more favorable with regards to angiogenesis process intensity, along with all its consequences and implications.

ELIGIBILITY:
Inclusion Criteria:

* cholelithiasis

Exclusion Criteria:

* symptoms of acute cholecystitis, diabetes, body mass indx above 36 kg/m2 and autoimmunological diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cholelithiasis and indications for surgical treatment; the median age of the patients included in the study was 48,5 and ranged from 18 to 70 years. The ratio of female to male patients was identical within each group and amounted 7:3.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-01; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
IL-6, IL-8, IL-10, VEGF-A, Endostatin serum levels before the laparoscopies and 6, 24, and 48 h afterwards | January 2006 - March 2006

CONTACTS AND LOCATIONS:
Overall Officials: Ryszard Maciejewski, Md, PhD, Study Chair — Medical University of Lublin
Locations (1):
- Medical University of Lublin, Lublin, Lublin Voivodeship, Poland